CLINICAL TRIAL: NCT00987376
Title: Comparison of Novel PET/CT Imaging Agents and MRS/MRI in Metastatic and High Risk Prostate Cancer: An Inter-SPORE Collaboration
Brief Title: Novel PET/CT Agents and MRS/MRI in Prostate CA and High Risk Prostate Cancer: An Inter-SPORE Collaboration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Val Lowe, Val J. Lowe, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8-03; CA91956-02
Record Dates: First submitted 2007-12-20; First posted 2009-09-30 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Prostate cancer patients
  Interventions: Device: Diagnostic Imaging: C11 choline PET; C11 acetate PET; and MRI Spectroscopy

INTERVENTIONS:
Device: Diagnostic Imaging: C11 choline PET; C11 acetate PET; and MRI Spectroscopy — C11 Choline, C11 Acetate PET and MRI

SUMMARY:
Prostate cancer imaging using traditional anatomic modalities including CT, MR, and ultrasound is limited. Improvement in current imaging modalities or development of new ones should be a priority in prostate cancer research. Optimal treatment varies considerably for patients with different staging characterizations and new imaging methods that more accurately stage patients could lead to more appropriate treatment. The objective of this study is to obtain preliminary, comparative data on new, promising imaging methods for prostate cancer. PET/CT imaging using 11C-choline,11C-acetate, and Y86 or 18F-Adenosylcobalamin and MRI spectroscopy (MRS) of prostate cancer will be compared. Direct comparison of these imaging methods has never been done and Mayo Clinic and Johns Hopkins are uniquely able to conduct such a trial as an inter-SPORE collaboration.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 years of age or older
* Patients who have completed staging CT and/or bone scan as part of their routine workup
* Patients with bulky metastatic prostate cancer who have 5 or more lesions suspicious for distant metastases as determined by routine CT and/or bone scans that are untreated by radiation

Exclusion Criteria:

* Patients who are less than 6 weeks post operative for Greenfield filter placement
* Patients with metallic surgical implants including pacemaker implants, cochlear implants, dentures held in place by magnets imbedded in the gums and aneurysm clips except those inserted at Mayo and only those inserted after October of 1994 and /or metal fragments in the body including metal fragments in the eyes

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Test accuracy | 2 years

SECONDARY OUTCOMES:
Test comparative accuracy of PET and MRI | 2years

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States